CLINICAL TRIAL: NCT03875794
Title: OMILQ: Osteopathic Manipulation to Increase Lactation Quantity (OMILQ)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There is no one to transfer to study to and no one interested in this research study. I am taking 8 months off from being a physician so the study needs to be closed
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1174025
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Osteopathic Manipulation
Keywords: Lactation; Insufficient, Partial; Lactating Female
MeSH Terms: conditions — Breast Feeding | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osteopathic Manipulation (Experimental): This research will be carried out as a prospective, non-randomized pilot study in women aged 18-40 who are 2 weeks to 28 weeks postpartum.
  The intervention investigated in this study is osteopathic manipulation.
  Interventions: Other: Osteopathic Manipulation

INTERVENTIONS:
Other: Osteopathic Manipulation — Using osteopathic manipulation as an intervention to increase milk supply in lactating women.

SUMMARY:
This study is designed to investigate whether using osteopathic manipulation can increase the milk supply in lactating women.

DETAILED DESCRIPTION:
The short and long-term benefits of breastfeeding to both the mother and infant are well established. Benefits for the child range from protection against common childhood infections, decreased rates of type-2 diabetes and systolic hypertension, lower rate of sudden infant death syndrome, increased performance on intelligence tests, and possible reduction in obesity. Maternal benefits include a reduction in the risk of breast cancer, diabetes, hyperlipidemia, hypertension, myocardial infarction, obesity, and ovarian cancer. Given this evidence the World Health Organization (WHO) and the American Academy of Pediatrics recommend, exclusive breastfeeding of infants for the first six months. WHO goes on to recommend breastfeeding to 2 years and beyond if mutually agreeable to both the mother and child. Despite these benefits and recommendations, according to the Centers for Disease Control and Prevention (CDC) in the United States 81% of infants were started breastfeeding and only 51% continued at 6 months. Perceived or actual low milk supply is one of the most common reasons for discontinuing breastfeeding.

This protocol is designed to investigate scientifically our current osteopathic standard of care. There is no available research data to date specifically on using osteopathic manipulation as an intervention to increase milk supply in lactating women.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 40
2. Between 2 and 28 weeks postpartum from a live infant birth weighing at least 2500g
3. Desire to exclusively breastfeed
4. Able to provide informed consent
5. Available for the duration of the study
6. 1 hour milk volume of less than 1oz (or 2oz for twins)
7. All current nurslings are the same age

Exclusion Criteria:

1. Current use of domperidone
2. Current use of metoclopramide
3. Current use of silymarin
4. History of breast surgery
5. Current malignancy
6. Current pulmonary embolism or deep vein thrombosis
7. Current medical condition resulting in increased intra-cranial pressure
8. History of insufficient glandular tissue (IGT)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Lactating females
Enrollment: 5 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
Lactation Volume | Baseline through 4 weeks
  Measuring lactation volume after osteopathic manipulation in ounces.

SECONDARY OUTCOMES:
Change in formula supplementation | Baseline to 4 weeks
  Change in lactation production in order to change the number of ounces needed for formula supplementation.
Change in reported self-worth | Baseline to 4 weeks
  Change in subject reported self-worth as assessed on an Investigator developed questionnaire (based off the Patient-Reported Outcomes Measurement Information System [PROMIS] questionnaire on a 5 point Likert scale).

CONTACTS AND LOCATIONS:
Overall Officials: Arlene O'Donnell, DO, Principal Investigator — AdventHealth
Locations (1):
- AdventHealth East Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No